CLINICAL TRIAL: NCT05158517
Title: VeDOlizumab PERsistence in IBD Patients After Switching From Intravenous to Subcutaneous Administration : a Real-life Multicenter Study
Brief Title: VeDOlizumab PERsistence in IBD Patients After Switching From Intravenous to Subcutaneous Administration : a Real-life Multicenter Study (DOPER)
Acronym: DOPER
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: GT-2021-04
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD UC
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Subcutaneous vedolizumab — Patients will be switched from IV vedolizumab into subcutaneous vedolizumab

SUMMARY:
Descriptive : A 12-months multicenter, observational, prospective cohort study. Population : IBD patients under stable clinical and biological remission will be proposed to switch from the IV vedolizumab to the SC vedolizumab as part of routine care. All consecutive IBD patients in IBD centers participating in the study will be proposed to participate in the study during their regular outpatients' visits.

Objectives : The primary objective of DOPER study is to describe SC vedolizumab persistence after switching from IV vedolizumab to SC vedolizumab at month 12.

DETAILED DESCRIPTION:
Number of patients : 400 patients in approximatively 31 sites in France. Recrutment period : The trial duration for each patient will be 1 year main. Endpoint : The primary endpoint is to assess the rate of persistence of SC vedolizumab at month 12 after switching from IV vedolizumab to SC vedolizumab.

Secondary Endpoint :

* Percentage of clinical remission at months 3 and 12, defined as a Partial Mayo Score (PMS) <2 with each sub-score (stool frequency, rectal bleeding, and physician rating of disease activity) of 1 or less for UC patients and as a Harvey Bradshaw Index (HBI) score ≤4 for CD patients
* Percentage of steroid free clinical remission at month 12
* Percentage of biological remission rates (defined as fecal calprotectin <250 μg/g and C-Reactive-Protein (CRP) <5 mg/L) at month 12
* Percentage of Patient-Reported Outcome 2 (PRO-2, defined as stool frequency and rectal bleeding for UC and stool frequency and abdominal pain for CD) response and remission at month 12
* Percentage of clinical relapse free rates at month 12
* Percentage of loss of response rates at month 12
* Mean change from baseline in PMS or HBI, CRP and fecal calprotectin compared to month 12
* Percentage of patients who switch back to previous IV vedolizumab therapy at month 12after switching from IV vedolizumab to SC vedolizumab
* Proportion of patients with positive antibodies (VDZ, ANA) comparing therapy with IV and SC vedolizumab
* Persistence of SC vedolizumab at month 12 in patients previously treated by IV vedolizumab every 4 weeks, compared to patients treated by IV vedolizumab every 8 weeks
* Twelve-month cumulative surgery rates
* Hospitalization rate at month 12
* Cumulative infection rate at month 12
* Cumulative injection reactions at month 12
* Cumulative adverse events (AEs) rate at month 12
* Comparison between incidence of specific anti-drug antibodies and incidence of AEs

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are more than 18 years of age, on the day of signing informed consent
* Documented diagnosis of IBD, established on the basis of standard clinical, endoscopic and/or histological criteria.
* CD or UC remission defined per clinical assessment as a Harvey Bradshaw Index (HBI) score ≤4 for CD patients and a Partial Mayo Score (PMS) < 2 with each sub-score of 1 or less for UC and/or according to ECCO classification within previous 3 months
* Currently treated with IV vedolizumab
* Patients agreeing to switch from IV to SC formulation
* Receiving or not the concomitant following drugs (but must remain on stable dose for 12 weeks):

  * Oral 5-aminosalicylates (5ASA) compounds or rectal formulations of 5ASA provided the dose to be stable at least 4 weeks before switching
  * Azathioprine, 6-Mercaptopurine or methotrexate provided the dose has been stable for 4 weeks prior to inclusion • Each patient is required to provide written informed consent in order to be included in the study

Exclusion Criteria:

* Current use of adalimumab, infliximab, golimumab or ustekinumab
* Current use of JAK inhibitors or S1P modulators
* Current use of steroids or within the last three months for IBD
* Treatment with any investigational agent in the past 30 days or five half-lives prior to the screening visit (whichever is longer)
* Active clinically significant infection or HIV, Hep B, Hep C, untreated tuberculosis
* Female subjects with pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years old, CD patients (HBI ≤ 4) or UC patients (PMS ≤ 2) with established diagnosis > 6 months treated with vedolizumab IV, agreeing to switch from IV to SC formulation or who have just switched to subcutaneous vedolizumab as part of routine care
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous vedolizumab dosage after switch | Month 12
  To describe subcutaneous vedolizumab persistence after the switch from IV vedolizumab to SC vedolizumab at month 12
Efficacy of subcutaneous vedolizumab treatment in clinical remission | Month 12
  Steroid-free clinical remission 12 months after switching
Safety of subcutaneous vedolizumab treatment | Month 12
  Proportion of participants with treatment-related adverse events for a period of 12 months after swiching

SECONDARY OUTCOMES:
Ratio efficacy of SC vedolizumab in clinical remission | Month 12
  Percentage of patients on steroid free clinical remission at month 12 after switch :
  Steroid-free Clinical remission is defined as a Partial Mayo Score (PMS) <2 with each sub-score (stool frequency, rectal bleeding, and physician rating of disease activity) of 1 or less for UC patients and as a Harvey Bradshaw Index (HBI) score ≤4 for CD patients
Loss of response to vedolizumab SC treatment | Month 12
  Percentage of patients who switch back to originator previous therapy IV vedolizumab at month 12 after switching from IV vedolizumab to SC vedolizumab in IBD patient
Efficacy of SC vedolizumab treatment on patient quality of life | Month 12
  Percentage of PRO2 response and remission at month 12
Efficacy of SC vedolizumab treatment in biological remission | Month 12
  Percentage of biological remission rates (FC<250μg/g, CRP<5mg/L) at month 12
Efficacy of SC vedolizumab treatment in preventing relapse | Month 12
  Percentage of clinical relapse free rates at month 12
Efficacy of SC vedolizumab treatment in preventing loss of response | Month 12
  Percentage of loss of response rates at month 12
Loss of clinical response | Month 3
  Percentage of clinical response and remission at month 3
Disease activity | Moth 12
  Mean change from baseline in :
  * For Crohn Disease : HBI (Harvey Bradshow Index)
  * For Ulcerative Colitis : PMS (Partiel Mayo Score)
  * Biological criteria : CRP (mg/L) : Remission < 5 mg CRP in 1 litre of blood and fecal calprotectin (μg/g) : remission < 250 μg of fecal calprotectin in 1g of stool HBI score, PMS score, CRP ad calprotectin fecal will be combined to report the disease activity (this outcome is expressed without units)
Treatment adherence | Month 12
  Proportion of patients with positive antibodies (VDZ, ANA) comparing therapy with original and SC vedolizumab
Medication Possession Ratio (MPR) | Month 12
  Adherence to biosimilar switch during the follow-up : MPR ratios

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Chateau, Grenoble, Auvergne-Rhône-Alpes, France